CLINICAL TRIAL: NCT03975309
Title: Metabolomics of Neurocognitive Risk for Dementia in Diabetes
Brief Title: DHS MIND Metabolomics
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00057194; 1R01AG058921-01A1 (NIH)
Record Dates: First submitted 2019-05-28; First posted 2019-06-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Diabetes
Keywords: Cognition, Dementia, Mild Cognitive Impairment, European American, African American
MeSH Terms: conditions — Diabetes Mellitus; Dementia; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, urine, blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Previous DHS Participants: Observational

SUMMARY:
The study team will evaluate whether metabolomic signatures of neurocognitive decline trajectories are exacerbated by the presence of type 2 diabetes mellitus (T2D) and whether these signatures contribute in part, to ethnic disparities in cognitive decline between European Americans and African Americans with T2D.

DETAILED DESCRIPTION:
Aim 1. Re-examine the Diabetes Heart Study Memory IN Diabetes (DHS MIND) cohort for progression of neurocognitive decline using an established cognitive battery, literacy testing, and adjudicated physician diagnosis of dementia.Another neurocognitive evaluation will be completed in European-American and African-American DHS MIND participants, providing longitudinal follow-up more than eight years after initial assessment. The cognitive battery will reassess domains of executive function, memory, and global cognition. In addition, a clinical exam will include a literacy evaluation to circumvent the shortcomings of differences in educational attainment among participants. A physician adjudicated assessment of cognitively normal, mild cognitive impairment, or dementia will be obtained. Cognitive evaluations will inform epidemiological analyses regarding cross-sectional and trajectories of cognition decline relative to existing and repeat measures of cardio-metabolic risk factors.

Aim 2. Examine the metabolomic basis of neurocognitive measures in people with T2D. The presence of T2D, cardiovascular disease and reduced kidney function are significant risk factors for development of cognitive impairment. These risk factors are enriched in the DHS and lack early diagnostic tools. Untargeted metabolomic profiling offers the potential to identify relevant biomarkers that could impact the diagnosis, prognosis, and treatment of cognitive decline. This will be accomplished through untargeted metabolomic analysis of European American and African American DHS MIND participants using stored samples from baseline visits acquired more than 10 years prior to the current (repeat) neurocognitive assessment. These data will be used to A) provide information on novel mechanistic insights into cognition and trajectories of cognitive decline, B) develop a risk prediction model using the baseline exam, and C) validate extremes of neurocognitive performance using longitudinal assessments while examining ancestry/ethnic-specific differences.

Aim 3. Comprehensive genetic analysis of DHS participants to examine the genetic architecture of metabolomic signatures associated with the trajectories of neurocognitive decline. Existing genome-wide data will be used to map regions of the human genome that contain loci contributing to measures of neurocognition and metabolomics signatures of change in these variables through longitudinal assessment. Causal effect modeling will validate the association of modifiable exposures, i.e. genetic markers and metabolites on the outcome (i.e. trajectories of neurocognitive decline).

ELIGIBILITY:
Inclusion Criteria:

• At the baseline visit, European American and African American individuals with T2D must have had diabetes diagnosed after the age of 30, 3 years disease duration and lack historical evidence of diabetic ketoacidosis.

Exclusion Criteria:

* At the baseline visit, participants with pre-existing kidney disease, defined as a serum creatinine concentration >1.5 mg/dl or blood urea nitrogen >35 mg/dl were excluded due to the elevation of serum AGE levels in individuals with kidney disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: European Americans and African Americans with T2D from the general population.
Sampling Method: Non-Probability Sample
Enrollment: 417 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Wide Range Achievement Test 4 (WRAT 4) | up to 25 years prior to Day 1
  Word reading subtest to measure letter and word decoding through word recognition and letter identification. This outcome is a data pull/chart review from a previous study for some of the participants.Score range is 0-70, 70 is the best score possible.
Wide Range Achievement Test 4 (WRAT 4) | Day 1
  Word reading subtest to measure letter and word decoding through word recognition and letter identification. Score range is 0-70, 70 is the best score possible.
Rey Auditory Verbal Learning Test (RAVLT) | up to 25 years prior to Day 1
  A word recall list that measures verbal learning and memory. Involves immediate and delayed recall. This outcome is a data pull/chart review from a previous study for some of the participants. Score range is 0-75, 75 is the best possible score.
Rey Auditory Verbal Learning Test (RAVLT) | Day 1
  A word recall list that measures verbal learning and memory. Involves immediate and delayed recall. Score range is 0-75, 75 is the best possible score.
Modified Mini-Mental State Exam (3MSE) | up to 25 years prior to Day 1
  Measures general cognitive function. This outcome is a data pull/chart review from a previous study for some of the participants. Score range is 0-100, 100 is the best possible score.
Modified Mini-Mental State Exam (3MSE) | Day 1
  Measures general cognitive function. Score range is 0-100, 100 is the best possible score.
Digit Symbol Coding Task (DSC) | up to 25 years prior to Day 1
  DSC is a subtest of the Wechsler Adult Intelligence Scale III or IV. It is used to access visual motor speed. This outcome is a data pull/chart review from a previous study for some of the participants. Score range 0-133, 133 is the best possible score.
Digit Symbol Coding Task (DSC) | Day 1
  DSC is a subtest of the Wechsler Adult Intelligence Scale III or IV. It is used to access visual motor speed. Score range 0-133, 133 is the best possible score.
Stroop subtests 1, 2 and 3 | up to 25 years prior to Day 1
  Measures executive function by determining interchanging word and color challenges. This outcome is a data pull/chart review from a previous study for some of the participants. Score range 0-420 seconds, the lower time point is the best.
Stroop subtests 1, 2 and 3 | Day 1
  Measures executive function by determining interchanging word and color challenges. Score range 0-420 seconds, the lower time point is the best.
Category Fluency for Animals | up to 25 years prior to Day 1
  Measures verbal fluency and language aspects of executive function by asking participant to name as many unique items as possible in a category ie. animals. This outcome is a data pull/chart review from a previous study for some of the participants. Score 0-26, the best possible score is 26.
Category Fluency for Animals | Day 1
  Measures verbal fluency and language aspects of executive function by asking participant to name as many unique items as possible in a category ie. animals. Score 0-26, the best possible score is 26.
Montreal Cognitive Assessments (MoCA) | up to 25 years prior to Day 1
  Measures general cognitive and executive function, has increased sensitivity for detecting early cognitive impairment.This outcome is a data pull/chart review from a previous study for some of the participants. Score range is 0-30, 30 is the best possible score.
Montreal Cognitive Assessments (MoCA) | Day 1
  Measures general cognitive and executive function, has increased sensitivity for detecting early cognitive impairment.Score range is 0-30, 30 is the best possible score.

SECONDARY OUTCOMES:
Craft Story Recall (Immediate/Delayed) | Day 1
  Assesses the ability to retell a story from memory immediately and after a delay of approximately 20 minutes. Score 0-69 (for each portions of the test). The best possible score is 69.
Trail Making Test | Day 1
  Measures processing speed and executive function. Part A- Score 0-150 sec, Part B Score 0-300 sec, the fastest time is better.
Number Span Test (Forward/Backward) | Day 1
  Assesses working memory recalling numbers said forwards and backwards in increasing number of digits. Score 0-28, the best score possible is 28.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholette D Allred, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No